CLINICAL TRIAL: NCT00692809
Title: Impact of HIV Infection on Latent TB Among Patients With HIV-TB Co-infection
Brief Title: Impact of HIV Infection on Latent Tuberculosis (TB) Among Patients With HIV-TB Co-infection
Acronym: HIV-TB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology, India (Other Government)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Dr. S.K. Sharma, Professor & Head, All India Institute of Medical Sciences
Other Study IDs: SKS/LTBI/07
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2008-06

CONDITIONS: Latent Tuberculosis Infection; HIV Infections; Tuberculosis
Keywords: Latent tuberculosis infection; Human immunodeficiency virus; Tuberculosis; Natural Killer T Cells; Invariant Natural Killer T Cells; Regulatory T cells; Interferon-gamma
MeSH Terms: conditions — Latent Tuberculosis; HIV Infections; Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: HIV+ve+LTBI (n=100)
- 2: HIV+ve+clinical TB (n=50)
- 3: HIV-ve+clinical TB (n=15)
- 4: Normal control (n=15)

SUMMARY:
HIV induced altered representation and function of regulatory T cell subsets (NKT and Treg cells) impair the protective T cell response against M.tuberculosis and disrupts LTBI, thus facilitates faster progression and development of severe forms of clinical TB in HIV-TB co-infection.

DETAILED DESCRIPTION:
During the natural course of HIV disease, emergence of opportunistic infection not only imposes morbidity on HIV-TB co-infected patients, but also facilitates viral replication causing faster disease progression. Tuberculosis, being the commonest among the opportunistic infections among HIV infected persons deserves special attention. Moreover, disruption of latency of TB infection (LTBI) with development of more severe clinical forms at relatively early stage of HIV disease when CD4 count still remains above 300/ul, makes TB a unique opportunistic infection and negatively influence the outcome of dual infection.This is suggestive of impairment of some critical immune function involving relatively less frequent fine T cell subsets with functional hierarchy over bulk T cells, so as to weaken the immune containment of LTBI resulting in reactivation of M. tuberculosis and manifestation of severe forms of TB.HIV has recently been reported to preferentially infect, destroy and incapacitate two key immune-regulatory T cell subsets, namely NKT and Treg cells.Therefore, studying them along the course of HIV disease and impact of their changes on the function of effector T cells directed against M.tuberculosis is important.

ELIGIBILITY:
Inclusion Criteria:

HIV infected +LTBI group:

* Patient of either sex between 18-65 years of age
* All the patients should be HIV ELISA test positive irrespective of CD4 count and presence of other opportunistic infections Antiretroviral drug naive HIV patients
* No past history of TB
* Patients should be either tuberculin test positive (> 5mm) or interferon gamma release assay positive
* Written informed consent to participate in the study given by participants or legal guardian
* Patients able to comply with instructions and come back for a regular follow up

HIV infected + Clinical TB group:

* Patient of either sex between 18-65 years of age
* All the patients should be HIV ELISA test positive irrespective of CD4 count and presence of other opportunistic infections
* In PTB group, patient should be two sputum smear positive out of three consecutive samples
* In EPTB group, diagnosis of TB will be:

  * Definitive -Culture confirmed
  * Probable -Histopathological or radiological -Clinical features and response to anti TB treatment (ATT)
  * Possible TB -Clinical feature and response to anti TB treatment (ATT)
* Written informed consent to participate in the study given by participants or legal guardian
* Patients able to comply with instructions and come back for a regular follow up

HIV negative Clinical TB group:

* Patients of either sex between 18-65 years of age who are permanent resident of Delhi
* All patients should be HIV ELISA negative
* In PTB group, patients should be two sputum smear positive (at least 1+) out of three consecutive samples
* In EPTB group, diagnosis of TB will be:

  * Definitive -Culture-confirmed
  * Probable -Histopathological or radiological -Clinical features and response to anti-TB treatment (ATT)
  * Possible TB -Clinical features and response to anti-TB treatment (ATT)
* Written informed consent to participate in the study given by participants or legal guardian
* Patients able to comply with instructions and come back for a regular follow up

Normal controls:

* Persons of either sex between 18-65 years of age who are permanent resident of Delhi
* Written informed consent to participate in the study given by participants or legal guardian
* Person should not have past history of TB

  * Mantoux test negative (< 10mm)
  * Chest-X-ray normal
  * Hemogram normal
* Renal and liver functions normal
* Hepatitis viral markers normal
* No clinical evidence of malnutrition
* HIV ELISA negative

Exclusion Criteria:

HIV infected +LTBI group:

* Pregnant and lactating females
* Patients who are getting steroid therapy
* Transplant patients, diabetes mellitus or malignancy, chronic renal failure or liver diseases
* Currently receiving cytotoxic therapy, or have received it within the last 3 months
* Terminally ill as per treating clinician's judgment
* Patient from outside Delhi and migrants

HIV infected + Clinical TB group:

* Category II and multidrug-resistant pulmonary tuberculosis
* Pregnant and lactating females
* Patients who are getting steroid therapy
* Transplant patients, diabetes mellitus or malignancy, chronic renal failure or liver diseases
* Currently receiving cytotoxic therapy, or have received it within the last 3 months
* Terminally ill patient as per treating clinician's judgment
* Patients from outside Delhi and migrants

HIV negative Clinical TB group:

* Category II and multi drug-resistant pulmonary tuberculosis
* Patients who are getting steroid therapy
* Transplant patients, diabetes mellitus or malignancy, chronic renal failure or liver disease
* Currently receiving cytotoxic therapy, or have received it within the last 3 months
* Terminally ill patient as per treating clinician's judgment
* Patients unwilling to comply with the study procedures or those with history of alcohol or drug abuse

Normal controls:

* Transplant patients, diabetes mellitus or malignancy
* Patients unwilling to comply with the study procedures or those with history of alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV+ve+LTBI HIV+ve+clinical TB HIV-ve+clinical TB Normal control
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Precise component(s) of T cell response against M.tuberculosis compromised by HIV infection which leads to the development of severe forms of clinical tuberculosis. | 5 months

SECONDARY OUTCOMES:
Elucidation of critical events of the cellular and molecular interactions that would be useful for developing newer therapeutic strategies and vaccination. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, M.D., Ph.D, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India